CLINICAL TRIAL: NCT00323245
Title: Regaining Urinary Continence in Postmenopausal Women With Osteoporosis: A Randomized Controlled Trial.
Brief Title: Regaining Bladder Control in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Meena Sran, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C05-0608; W05-0259
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Urinary Incontinence
Keywords: Randomized clinical trial; osteoporosis; urinary incontinence; physiotherapy; education
MeSH Terms: conditions — Urinary Incontinence; Osteoporosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Physiotherapy for urinary incontinence — See Detailed Description.

SUMMARY:
Conservative management for urinary incontinence has been shown to improve bladder control. We are conducting a study of the effectiveness of conservative management for urinary incontinence in women who also have osteoporosis. We hope to find that treatment for incontinence improves bladder control and thereby allows women to be more active and reduces their risk of falling and breaking bones.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women osteopenia or osteoporosis and stress urinary incontinence

Exclusion Criteria:

-

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Number of Incontinent Episodes (baseline and end of treatment (12 weeks)

SECONDARY OUTCOMES:
Urinary Distress Inventory
Pelvic Floor Muscle Strength
Quality of life: Each participant will complete the Incontinence Impact Questionnaire and the SF-36 at the initial and follow up measurement sessions
Physical Activity (PASE)
24 Hour Pad Test
Voiding Frequency using the bladder diary
Spinal Curvature with a flexicurve ruler
Self-Perceived Efficacy
All at initial and follow up (end) measurement sessions

CONTACTS AND LOCATIONS:
Overall Officials: Meena Sran, PT, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- BC Womens' Health Centre, Vancouver, British Columbia, Canada